CLINICAL TRIAL: NCT06605833
Title: CARD-IO - CARDiac Toxicity Following ImmunOtherapy Treatment for Melanoma
Brief Title: CARDiac Toxicity Following ImmunOtherapy Treatment for Melanoma
Acronym: CARD-IO
Status: Enrolling by invitation | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR6063
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Melanoma Stage III or IV
Keywords: melanoma; cardiac toxicity; immune related adverse events; immunotherapy treatment
MeSH Terms: conditions — Melanoma; Cardiotoxicity | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 2-4 years: Patients on routine follow-up 2-4 years after the completion of immunotherapy treatment for melanoma
  Interventions: Diagnostic Test: 12-Lead ECG; Diagnostic Test: Transthoracic Echocardiogram; Diagnostic Test: Cardiac MRI; Diagnostic Test: Cardiac Biomarker Screening; Other: Basic Observations
- 5-7: Patients on routine follow-up 5-7 years after the completion of immunotherapy treatment for melanoma
  Interventions: Diagnostic Test: 12-Lead ECG; Diagnostic Test: Transthoracic Echocardiogram; Diagnostic Test: Cardiac MRI; Diagnostic Test: Cardiac Biomarker Screening; Other: Basic Observations
- 8-10+: Patients on routine follow-up 8-10+ years after the completion of immunotherapy treatment for melanoma
  Interventions: Diagnostic Test: 12-Lead ECG; Diagnostic Test: Transthoracic Echocardiogram; Diagnostic Test: Cardiac MRI; Diagnostic Test: Cardiac Biomarker Screening; Other: Basic Observations

INTERVENTIONS:
Diagnostic Test: 12-Lead ECG — Participants will undergo a standard 12-lead ECG in order to record the electrical activity of the heart. This typically takes a few minutes and the ECG is read by a cardiologist
  This is a Standard of Care test being performed at a non Standard of Care timepoint
Diagnostic Test: Transthoracic Echocardiogram — A transthoracic echocardiogram will be performed in accordance to standard British Society of Echocardiography guidelines. This will involve undertaking an ultrasound scan of the participant's heart with ultrasound jelly to obtain information including left ventricular function and valvular function.
  This is a Standard of Care test being performed at a non Standard of Care timepoint
Diagnostic Test: Cardiac MRI — A cardiac MRI scan will be performed in order to assess the morphology and function of the heart in accordance with international guidelines. Data that will be derived includes biventricular volumes and function and myocardial strain data.
  This is a Standard of Care test being performed at a non Standard of Care timepoint
Diagnostic Test: Cardiac Biomarker Screening — * Cardiac Troponin I,
  * NTproBNP],
  * lipid profile,
  * HbA1c
  * ferritin
  These are Standard of Care tests being performed at a non Standard of Care timepoint
Other: Basic Observations — * Heart rate
  * Blood pressure
  * Oxygen SAT
  * Respiratory rate
  These are Standard of Care observations being performed at a non Standard of Care timepoint

SUMMARY:
People who develop a type of skin cancer known as 'melanoma' are often treated with immunotherapy. The type of immunotherapy used for patients with melanoma is known as Immune Checkpoint Inhibitors (ICI). While ICI is very successful, it can lead to negative side effects that are known as 'immune related adverse events' (irAEs). These irAEs can affect any part of the body and can range in severity from mild symptoms to death.

There has been a lot of research on irAEs that occur during ICI, but less is known about how irAEs can affect people in the long-term.

Although irAEs are common from ICI, acute irAEs affecting the heart (cardiac irAEs) are uncommon. However, as they relate to the heart, they are often serious and have a higher rate of death compared to other types of irAEs. Little is known regarding the long-term effects of ICI on the heart. However, there is some evidence to suggest that ICI may also cause long-term cardiac irAEs such as accelerating a build-up of fatty materials in the arteries known as 'atherosclerosis' and inflammation of plaque in the heart. This can lead to an increased risk of heart attack.

Although there are guidelines for patients on ICI treatment to receive investigations to look for irAEs, including cardiac irAEs, there are no guidelines for monitoring long-term survivors.

The aim of the CARD-IO study is to establish if it is possible to investigate in long-term follow-up cardiac side-effects in patients who received ICI for melanoma. The data for this study would be used to support a larger study in the same patient population. Potentially, this could lead to a change in guidelines and long-term follow-up care for melanoma patients who have received ICI.

DETAILED DESCRIPTION:
Primary aim • To establish the feasibility of conducting a study to investigate late cardiac side effects caused by immunotherapy in patients with melanoma in order to generate data to support a larger study in this patient population.

Secondary aims

* To assess factors impacting on the acceptance and adherence with cardiac investigations.
* To contribute to the understanding of long-term cardiac toxicities following immunotherapy which will enable their early recognition.

Primary endpoint

• Acceptance rate (reported as the total number of patients consented divided by the number of patients invited for the study).

Secondary endpoints

* Adherence rate (reported as the proportion of patients completing all the scheduled cardiac screening tests divided by the number of patients enrolled in the study).
* Recruitment rate (reported as the number of patients recruited on average per month in each site, and overall).
* Reasons for non-adherence or declining to consent.
* Difference in adherence rates between adjuvant early disease setting and metastatic setting.
* Proportion of patients who experience cardiac irAEs during long-term follow-up, post-treatment.
* Prevalence of cardiac irAEs.

The planned sample size is 60 participants.

The project will assess 3 groups of patients at different timepoints during their standard of care surveillance, at 2-4, 5-7 and 8-10 years following the completion of their immunotherapy treatment for melanoma. Patients on routine follow-up, at 2 to 10 years following the completion of immunotherapy treatment for melanoma will be identified by searching through database of patients with melanoma who received immune checkpoint inhibitors (ICI). Patients respecting the inclusion criteria will be invited to take to part to the study.

Patients included in the study will undergo screening blood tests including cardiac biomarkers (troponin I, NTproBNP, lipid profile, HbA1c, ferritin), a 12 lead ECG and transthoracic echocardiography, a cardiac MRI alongside completing a questionnaire about cardiac events and risk factors. Patients will have blood tests done at Royal Marsden or Royal Free, while all the other cardiac investigations (ECG, transthoracic echocardiography, cardiac MRI) will be performed at the Royal Brompton Hospital. Surveillance imaging performed as per standard of care at the Royal Marsden or at the Royal Free will be reviewed for evidence of atherosclerosis by the team at the Royal Brompton. The cardiology team at the Royal Brompton will review cardiac investigations' results and abnormal results will be flagged.

A summary report will be generated and sent to the patients, their GPs, and the Site irrespective of the results found, and abnormal results will be investigated as per standard of care. The prevalence of cardiac adverse events will be summarised.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18 years or older
* Confirmed diagnosis of melanoma
* Stage IIB or IIC or stage III or stage IV melanoma
* Previous immunotherapy with immune-checkpoint inhibitors (anti PD-(L)1 +/- anti CTLA-4) for melanoma
* On standard of care surveillance, at 2 to 10+ years following the completion of immunotherapy treatment

Exclusion Criteria:

* Medical or psychological condition that would preclude informed consent.
* Known contraindications to MRI, such as claustrophobia, pregnancy, or indwelling metallic implant which is not MR conditional
* Current active treatment with systemic therapy for any malignancy.
* Active treatment with systemic therapy for any malignancy started after the completion of immunotherapy for melanoma.
* Subjects unable to comply with the study or sample schedule.
* Planned participation in a drug trial receiving investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from The Royal Marsden NHS Foundation Trust (RMH) and the Royal Free London NHS Trust (RFH) who are in follow up after receiving immunotherapy for melanoma 2-10+ years prior to enrolment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Acceptance rate | 12 months
  total number of patients consented divided by the number of patients invited for the study

SECONDARY OUTCOMES:
Adherence rate | 12 months
  proportion of patients completing all the scheduled cardiac screening tests divided by the number of patients enrolled in the study
Recruitment rate | 12 months
  Number of patients recruited on average per month in each site, and overall
Reasons for non-adherence or declining to consent | 12 months
  Reasons for non-adherence or declining to consent
Difference in adherence rates | 12 months
  Difference in adherence rates between adjuvant early disease setting and metastatic setting
Proportion of patients who experience cardiovascular irAEs | 12 months
  Proportion of patients who experience cardiovascular irAEs during long-term follow-up, post-treatment
Prevalence of cardiac irAEs | 12 months
  Prevalence of cardiac irAEs

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study to support the application of a larger more complex study by the same team on the same topic. Sharing of IPD would require additional consents and level of complexity in the Data Plan which current resource restraints does not allow. This will be considered for future studies based on this research.